CLINICAL TRIAL: NCT05554601
Title: A Randomized Trial of Behaviorally Designed Gamification and Social Incentives to Increase Physical Activity Among Overweight and Obese Veterans
Acronym: STEP 4 Vets
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 20-120
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Obesity
Keywords: physical activity
MeSH Terms: conditions — Hypertension; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: behavioral economics approach (gamification with social incentives)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- attention control (No Intervention): participants receive a FitBit and set goals but do no other intervention
- gamification with collaboration (Experimental): participants receive a FitBit and set goals, then are assigned to a group of other participants who will play a game to gain points based on collaboration with each other
  Interventions: Behavioral: gamification with collaboration
- gamification with competition (Experimental): participants receive a FitBit and set goals, then are assigned to a group of other participants who will play a game to gain points based on competition with each other
  Interventions: Behavioral: gamification with competition

INTERVENTIONS:
Behavioral: gamification with collaboration — participants receive a FitBit and set goals, then are assigned to a group of other participants who will play a game to gain points based on collaboration
  Arms: gamification with collaboration
Behavioral: gamification with competition — participants receive a FitBit and set goals, then are assigned to a group of other participants who will play a game to gain points based on competition with each other
  Arms: gamification with competition

SUMMARY:
Despite the many associated health benefits, more than half of Veterans do not achieve enough regular physical activity. The investigators' prior work has demonstrated that gamification, a method commonly used for health promotion, can lead to sustained increases in physical activity if it is designed using insights from behavioral economics to enhance social incentives. In this study, the investigators will compare the effectiveness of behaviorally designed gamification that encourages Veterans to collaborate or compete on physical activity levels and examine clinical outcomes as well as costs, barriers and facilitators to implementation of the program within Veterans Affairs.

DETAILED DESCRIPTION:
Background: Gamification is the use of game design elements such as points and levels in non-game contexts. Gamification is used commonly within workplace wellness programs and digital health applications; however, its effectiveness has been limited. A significant opportunity is to incorporate principles from behavioral economics, which have been effective in informing intervention designs that achieve sustained improvements in health behavior by addressing the 'predictable irrationality' of humans. The investigators' group has conducted two successful clinical trials using gamification and either collaboration or competition to increase physical activity in other settings. The investigators have conducted three pilot studies with Veterans to tailor these approaches to their specific needs and experiences.

Significance: Higher levels of regular physical activity are associated with reduced risk of cardiovascular disease, diabetes, hypertension, obesity, and mortality. Despite this, more than half of Veterans do not achieve enough physical activity to obtain these benefits.

Innovation and Impact: This will be one of the first clinical trials to incorporate behavioral economic principles and social incentives within the design of gamification to increase physical activity among obese Veterans with hypertension. It will also be one of the first to directly examine the impact of these interventions on clinical outcomes associated with increased physical activity and examine cost-effectiveness To improve scalability and decrease burden on Veterans, the entire study will be conducted completed remotely including enrollment and interventions. Moreover, the investigators will use state-of-the-art statistical and machine learning techniques to examine personalization of interventions.

Specific Aims: Aim 1: To evaluate the effectiveness of gamification with collaboration or competition to increase physical activity . Aim 2: To evaluate the effectiveness of gamification to improve clinical outcomes. Aim 3: To conduct a qualitative process evaluation and implementation analysis to inform implementation efforts within VA. Aim 4: To conduct a quantitative evaluation of Veteran characteristics related to demographics, past experiences, social networks, and other factors to identify heterogeneity in treatment effects. Aim 5: To assess the cost-effectiveness of the gamification interventions.

Methodology: Obese Veterans with hypertension will be enrolled into a three-arm randomized, controlled trial comprised of a 6-month intervention and a 3-month follow-up. Wearable devices will be used to passively monitor physical activity levels. Clinical outcomes will be captured by digital weight scales and blood pressure cuffs through video conferencing. Interventions will be deployed using Way to Health, a technology platform that the investigators have demonstrated is feasible to use within the VA Health System. Outcomes will include physical activity in steps (primary), minutes of moderate-to-vigorous physical activity (secondary), changes in clinical outcomes of weight and systolic blood pressure (secondary), change in minutes of sleep (exploratory), and cost of implementation (exploratory).

Next Steps/Implementation: The implementation analysis, which includes cost-effectiveness analysis and qualitative interviews with Veterans and key VA stakeholders, will inform implementation of the program in VA. The investigators have support from the following three operational partners to implement key learnings into existing VA programs: VA National Center for Health Promotion and Disease Prevention including MOVE!, VA Office of Connected Care, and the VA Chief Improvement and Analytics Officer.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care at the CMCVAMC age 18 or older with a body mass index > 30
* a hypertension diagnosis with systolic blood pressure >140mm Hg
* are interested in participating in a 9-month physical activity program

Exclusion Criteria:

* currently participating in another physical activity research study
* any medical conditions prohibiting ambulation without assistance
* if a 9-month physical activity program is infeasible or unsafe
* if the Veteran is at a higher level of physical activity (i.e., baseline step count >7500 steps per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
change in physical activity | 6 months
  change in mean steps per day from baseline to end of intervention

SECONDARY OUTCOMES:
blood pressure | 6 months
  change in systolic blood pressure from baseline to end of the intervention
weight | 6 months
  change in weight from baseline to end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Greysen, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA; Amol S. Navathe, MD PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waddell KJ, Patel MS, Clark K, Harrington TO, Greysen SR. Effect of Gamification With Social Incentives on Daily Steps After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2022 May 1;79(5):528-530. doi: 10.1001/jamaneurol.2022.0231. PMID 35344027
- [Background] Greysen SR, Waddell KJ, Patel MS. Exploring Wearables to Focus on the "Sweet Spot" of Physical Activity and Sleep After Hospitalization: Secondary Analysis. JMIR Mhealth Uhealth. 2022 Apr 27;10(4):e30089. doi: 10.2196/30089. PMID 35476034
- [Background] Largent EA, Eriksen W, Barg FK, Greysen SR, Halpern SD. Participants' Perspectives on Payment for Research Participation: A Qualitative Study. Ethics Hum Res. 2022 Nov;44(6):14-22. doi: 10.1002/eahr.500147. PMID 36316972

DOCUMENTS (1):
  • Informed Consent Form (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT05554601/ICF_000.pdf